CLINICAL TRIAL: NCT06113965
Title: Neural Operant Conditioning to Improve Walking After Stroke
Brief Title: Neural Operant Conditioning
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects enrolled
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, James Sulzer, James Sulzer, PhD, MetroHealth Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StudyID00000301
Record Dates: First submitted 2023-10-23; First posted 2023-11-02 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Chronic Stroke; Gait, Hemiplegic; Gait, Spastic; Walking, Difficulty
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic; Mobility Limitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Post-stroke Stiff-Knee Gait Participants (Experimental): Individuals with post-stroke Stiff-Knee gait
  Interventions: Device: Peripheral Nerve Stimulation

INTERVENTIONS:
Device: Peripheral Nerve Stimulation — Electrical stimulation of peripheral nerves to measure resulting gait kinematics and surface muscle activity

SUMMARY:
The goal of this clinical trial is to learn if operant conditioning can reduce spasticity in order to improve walking in stroke patient. The main questions it aims to answer are:

* Can participants self-regulate reflex excitability
* Can participants self-regulate reflex, reduce spasticity and improve walking Participants will undergo surface stimulation to evoke spinal reflexes and will be asked to control these reflexes therefore reducing spasticity.

Researchers will compare result to able bodied participants to see if [insert effects]

DETAILED DESCRIPTION:
The study purpose is to investigate the possibility and later effect of spinal reflex self-regulation in post-stroke stiff-knee gait. The intervention will consist of direct current surface stimulation of the peripheral nerves using electrical stimulation. Stimulation will evoke a motor response that will be collected through surface EMG electrodes and processed to depict a measure of the response as feedback to the participant to complete the loop of operant conditioning. The participant will attempt to modulate their responses over multiple sessions to cause this depiction to either increase or decrease its value depending on an established target.

.

ELIGIBILITY:
Inclusion Criteria:

1. Sign and date consent form
2. At least 3 months since stroke event
3. Over 18 years of age at time of eligibility
4. Ability to stand upright and walk for at least 5 minutes
5. Premorbidly independent
6. Mild to moderate gait impairment
7. Reduced knee flexion during walking relative to the unimpaired side
8. Unilateral hemiparesis of the lower limbs
9. Ability to evoke muscle responses through peripheral nerve stimulation, spinal cord stimulation, and transcranial magnetic stimulation
10. Medically stable
11. Skin intact on hemiparetic leg, abdomen, and scalp
12. Ability to evoke muscle responses and/or reflex responses through peripheral nerve stimulation, spinal cord stimulation, and/or transcranial magnetic stimulation

Exclusion Criteria:

1. Co-existing neurological condition other than prior stroke involving the hemiparetic lower limb (e.g., peripheral nerve injury, PD, SCI, TBI, MS).
2. History of lower limb musculoskeletal injury
3. Functionally relevant osteoarthritis and weight bearing restriction
4. Functionally relevant polyneuropathy resulting in lack of sensation in the lower leg
5. Functionally relevant cognitive impairment
6. Functionally relevant vision impairment
7. Pregnant
8. Botox injection to the ipsilateral leg in the last 12 weeks or taking oral anti-spasticity medications
9. Taking part in physical therapy for any walking-related impairment
10. Cardiac pacemaker or other implanted electronic systems
11. Uncontrolled seizure disorder
12. Use of seizure lowering threshold medications and the discretion of the study physician
13. Deficits in communication that interfere with reasonable study participation
14. Severely impaired cognition and communication
15. Severe lower limb pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Surface electromyographic recording of leg muscles | baseline, week 6 -mid-treatment, week 12 - end of treatment, 4-week post treatment, 12 weeks post treatment, 24 weeks post treatment
  Recording electrical activity of leg muscles during walking in response to peripheral nerve stimulation

SECONDARY OUTCOMES:
10 meter walk test | baseline, week 6 -mid-treatment, week 12 - end of treatment, 4-week post treatment, 12 weeks post treatment, 24 weeks post treatment
  10 meter walk test with collection of gait kinematics captured using an inertial motion capture camera system
quadriceps pendulum test | baseline, week 6 -mid-treatment, week 12 - end of treatment, 4-week post treatment, 12 weeks post treatment, 24 weeks post treatment
  This is a method of evaluating spasticity using gravity to provoke the muscular stretch reflex allowing for the collection of joint angle data. This data will aid in assessing changes in joint angles as a result of training.
Five Times Sit to Stand Test | baseline, week 6 -mid-treatment, week 12 - end of treatment, 4-week post treatment, 12 weeks post treatment, 24 weeks post treatment
  measures lower extremity functional strength. This test will measure your leg strength by asking you to sit down and stand up from a chair 5 times as fast as possible.
Transcranial Magnetic Stimulation (TMS) | Baseline, Week 12 - end of treatment
  non-invasive brain stimulation device, will be used to elicit a motor evoked response in participants via low frequency stimulation to the cortical regions associated with the muscles being investigated. This approach will test the integrity of the participant's CST in relation to the intervention and assessments being conducted

CONTACTS AND LOCATIONS:
Overall Officials: James Sulzer, PhD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Burpee JL, Lewek MD. Biomechanical gait characteristics of naturally occurring unsuccessful foot clearance during swing in individuals with chronic stroke. Clin Biomech (Bristol). 2015 Dec;30(10):1102-7. doi: 10.1016/j.clinbiomech.2015.08.018. Epub 2015 Sep 2. PMID 26371855
- [Background] Akbas T, Kim K, Doyle K, Manella K, Lee R, Spicer P, Knikou M, Sulzer J. Rectus femoris hyperreflexia contributes to Stiff-Knee gait after stroke. J Neuroeng Rehabil. 2020 Aug 26;17(1):117. doi: 10.1186/s12984-020-00724-z. PMID 32843057
- [Background] Li S, Francisco GE. New insights into the pathophysiology of post-stroke spasticity. Front Hum Neurosci. 2015 Apr 10;9:192. doi: 10.3389/fnhum.2015.00192. eCollection 2015. PMID 25914638
- [Background] Li S, Francisco GE, Zhou P. Post-stroke Hemiplegic Gait: New Perspective and Insights. Front Physiol. 2018 Aug 2;9:1021. doi: 10.3389/fphys.2018.01021. eCollection 2018. PMID 30127749
- [Background] Stoquart GG, Detrembleur C, Palumbo S, Deltombe T, Lejeune TM. Effect of botulinum toxin injection in the rectus femoris on stiff-knee gait in people with stroke: a prospective observational study. Arch Phys Med Rehabil. 2008 Jan;89(1):56-61. doi: 10.1016/j.apmr.2007.08.131. PMID 18164331
- [Background] Dehnadi Moghadam A, Hasanzadeh H, Dehnadi Moghadam F. Evaluation of the Effect of Intranasal Lidocaine in the Treatment of Spasticity in Patients with Traumatic Brain Injury. Anesth Pain Med. 2021 Aug 15;11(4):e115849. doi: 10.5812/aapm.115849. eCollection 2021 Aug. PMID 34692437
- [Background] Navarrete-Opazo AA, Gonzalez W, Nahuelhual P. Effectiveness of Oral Baclofen in the Treatment of Spasticity in Children and Adolescents With Cerebral Palsy. Arch Phys Med Rehabil. 2016 Apr;97(4):604-618. doi: 10.1016/j.apmr.2015.08.417. Epub 2015 Aug 28. PMID 26321489
- [Background] Wolpaw JR, Braitman DJ, Seegal RF. Adaptive plasticity in primate spinal stretch reflex: initial development. J Neurophysiol. 1983 Dec;50(6):1296-311. doi: 10.1152/jn.1983.50.6.1296. PMID 6663327
- [Background] Wolpaw JR, Lee CL. Motoneuron response to dorsal root stimulation in anesthetized monkeys after spinal cord transection. Exp Brain Res. 1987;68(2):428-33. doi: 10.1007/BF00248809. PMID 3480233
- [Background] Chen XY, Wolpaw JR. Operant conditioning of H-reflex in freely moving rats. J Neurophysiol. 1995 Jan;73(1):411-5. doi: 10.1152/jn.1995.73.1.411. PMID 7714584
- [Background] Thompson AK, Chen XY, Wolpaw JR. Acquisition of a simple motor skill: task-dependent adaptation plus long-term change in the human soleus H-reflex. J Neurosci. 2009 May 6;29(18):5784-92. doi: 10.1523/JNEUROSCI.4326-08.2009. PMID 19420246